CLINICAL TRIAL: NCT04807062
Title: Structural Bicortical Autologous Iliac Crest Bone Graft Combined With Tunnel Bone Tamps Method for Depressed Tibial Plateau Fractures
Brief Title: Treatment of Tibial Plateau Fractures With Bone-graft and Bone Tamp Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICBG001
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Depressed Tibial Plateau Fractures
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DTPFs treated with structural bicortical autologous ICBG combined with TBTM (Experimental)
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — tunnel bone tamps method (TBTM) was used to reduce the depressed articular fragments and then structural bicortical autologous ICBG was used to fill the valley tunnel.
  Other Names: Structural bicortical autologous iliac crest bone graft combined with tunnel bone tamps method

SUMMARY:
Autologous ICBG and bone tamp methods are often applied to manage depressed tibial plateau fracture (DTPF), but previous iliac bone harvesting and bone tamp techniques remain controversial. The purpose of this study is to describe and evaluate the technique of using structural bicortical autologous iliac crest bone-graft (ICBG) combined with tunnel bone tamps method (TBTM) in treating DTPFs.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age ≥ 18 years);
* diagnosis of DTPFs;
* agreeing to receive structural bicortical autologous ICBG combined with TBTM treatment and subsequent internal fixation treatment;
* agreeing to participate in regular follow-up after surgery.

Exclusion Criteria:

* open fracture;
* pathologic fractures;
* bone metabolic disease;
* previous ICBG;
* infection or soft tissue injury of the iliac bone donor site;
* pelvic fractures or bone tumors;
* associated peripheral nerve injury;
* non-completion of 30 months follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative immediate reduction rate | up to 2 weeks
  Preoperative and postoperative imaging data of all subjects, including X-ray and CT scans, were collected. Picture Archiving and Communication Systems (PACS) was used to measure articular step-off and evaluate the immediate reduction after surgery.
Postoperative long-term reduction rate | up to 2 weeks
  The immediate postoperative and follow-up imaging data of all subjects, including X-ray and CT scan, were collected. PACS system was used to measure the articular step-off and evaluate the long-term reduction after surgery.
Bone healing time | up to 2 weeks
  Postoperative follow-up imaging data of all patients were collected, including X-ray and CT scans.Evaluating the bone healing time based on callus growth.

SECONDARY OUTCOMES:
operative time | up to 1 weeks
  The operation time in the bone graft donor site and bone graft site of all subjects was recorded as the basis for evaluating the size of surgical trauma.
intraoperative blood loss | up to 1 weeks
  The intraoperative blood loss in the bone graft donor site and bone graft site of all subjects was recorded as the basis for evaluating the size of surgical trauma.
The incidence of complications in the bone-graft donor and bone-graft sites | up to 1 weeks
  Surging-related complications of all subjects were recorded as a basis for evaluating surgical outcomes.
the Visual Analog Scale scores of ICBG donor and bone-graft sites | up to 1 week
  The Visual Analog Scale pain scores (ranged from 0 to 10, 0 representing no pain and 10 representing maximal imaginable pain) of all subjects during postoperative follow-up were recorded as the basis for evaluating the surgical effect.
Hospital for Special Surgery score of knee | uo to 1 week
  The knee Hospital for Special Surgery scores (ranged from 0 to 100, 0 representing poor knee function and 100 representing normal knee function) of all subjects during the postoperative follow-up was recorded as the basis for evaluating the surgical effect.
36-Item Short-Form Health Survey score | up to 1 week
  36-Item Short-Form Health Survey scores (ranged from 0 to 100, 0 representing poor health and 100 representing normal health) of all subjects during postoperative follow-up were recorded as the basis for evaluating the surgical effect.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wei, Doctor, Principal Investigator — Hebei Medical University Third Hospital
Locations (1):
- the Third Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes
Structural bicortical autologous iliac crest bone graft combined with tunnel bone tamps method for depressed tibial plateau fractures
Supporting Information: Study Protocol
Time Frame: 2 years after the experiment was conducted
Access Criteria: all authors focusing on tibial plateau fractures

REFERENCES:
- [Result] Wang Z, Tian S, Zhao K, Zhang R, Yin Y, Zhu Y, Hou Z, Zhang Y. Neutrophil to lymphocyte ratio and fracture severity in young and middle-aged patients with tibial plateau fractures. Int Orthop. 2020 Dec;44(12):2769-2777. doi: 10.1007/s00264-020-04793-6. Epub 2020 Sep 8. PMID 32897401
- [Result] Luo CF, Sun H, Zhang B, Zeng BF. Three-column fixation for complex tibial plateau fractures. J Orthop Trauma. 2010 Nov;24(11):683-92. doi: 10.1097/BOT.0b013e3181d436f3. PMID 20881634
- [Result] Greimel F, Weber M, Renkawitz T, Voellner F, Freude T, Grifka J, Craiovan B. Minimally invasive treatment of tibial plateau depression fractures using balloon tibioplasty: Clinical outcome and absorption of bioabsorbable calcium phosphate cement. J Orthop Surg (Hong Kong). 2020 Jan-Apr;28(1):2309499020908721. doi: 10.1177/2309499020908721. PMID 32131684
- [Result] Myeroff C, Archdeacon M. Autogenous bone graft: donor sites and techniques. J Bone Joint Surg Am. 2011 Dec 7;93(23):2227-36. doi: 10.2106/JBJS.J.01513. PMID 22159859
- [Result] Adams D, Patel JN, Tyagi V, Yoon RS, Liporace F. A simple method for bone graft insertion during Schatzker II and III plateau fixation. Knee Surg Sports Traumatol Arthrosc. 2019 Mar;27(3):850-853. doi: 10.1007/s00167-018-5134-9. Epub 2018 Sep 12. PMID 30206655
- [Derived] Li Y, Yang S, Yang H, Lian X, Hou Z. Drain versus no-drain at the donor sites of iliac crest bone graft: a retrospective study. J Orthop Surg Res. 2024 Oct 21;19(1):675. doi: 10.1186/s13018-024-05147-3. PMID 39428517